CLINICAL TRIAL: NCT02176031
Title: Phase II Trial of Natalizumab (Tysabri®) Plus Prednisone for Initial Therapy of Acute Graft Versus Host Disease (aGVHD) of the Gastrointestinal Tract
Brief Title: Phase II Trial of Natalizumab + Prednisone for Initial Therapy of Acute GI GVHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Corey S. Cutler, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-140
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Graft Versus Host Disease
Keywords: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Natalizumab; Methylprednisolone; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Natalizumab (Experimental): Natalizumab-
  * (Day 0 and 28) Fixed dose Intravenous infusion over one hour. 2 hours observation completion of the infusion
  * At 4 weeks, if there has been less than a complete response participants can be treated with a second dose of natalizumab.
  * If participants have no response after one dose, they will be not be given a second dose.
  * Participants who receive a second dose of natalizumab will be evaluated for response at day 56 after first treatment dose administered.
  * Participants will be assessed for response to therapy with natalizumab at day +28, day +56, day +100, day + 180, and day +365.
  * Commercial supplies of Methylprednisolone (or equivalent steroid) will be utilized. The formulation, preparation and route of administration will be as per package insert
  Interventions: Drug: Natalizumab; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Natalizumab
  Other Names: Tysabri®
Drug: Methylprednisolone
  Other Names: Steroid

SUMMARY:
This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational drug Natalizumab in treating Acute Graft-Versus-Host Disease (GVHD) in the Gastrointestinal (GI) Tract.

DETAILED DESCRIPTION:
Natalizumab is a drug that was initially discovered as a treatment for autoimmune conditions. Natalizumab has been approved for use in patients with Multiple Sclerosis and Crohn's disease. In these diseases, the drug works to inhibit dysfunctional immune cells that are responsible for the symptoms seen in these diseases. Acute graft versus host disease is caused by a similar dysfunction of immune cells; Natalizumab is thought to inhibit these immune cells, similarly to how it does in Multiple Sclerosis and Crohn's disease. In this research study,the investigators are looking to see whether Natalizumab provides additional benefit to patients receiving standard treatment for acute graft versus host disease of the gastrointestinal tract.

Participants who fulfill eligibility criteria will be entered into the trial to receive Natalizumab.

* Participant will receive a dose of the natalizumab through intravenous infusion. Participants may receive a second dose at Day 28 if they experience a partial response or very good partial response.
* Scheduled Physical Examination at screening, during the week of first dose and at 28 days, 56 days, 100 days, 180 days and one year.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Participants must have acute Graft-Versus-Host Disease (GVHD) of the lower gastrointestinal tract as defined by the clinical impression of the treating physician, requiring systemic treatment. Minimum criteria for GI GVHD includes diarrhea of greater than 500 mL/day. Biopsy of the GI tract is required for study entry and must confirm the diagnosis of acute GVHD. Stool samples to rule out infectious causes of diarrhea, including norovirus, Clostridium difficile and other clinically indicated infections must also be negative. Eligibility includes:
* Acute GVHD developing after allogeneic hematopoietic stem cell transplantation (HSCT) using bone marrow, peripheral blood stem cells, or umbilical cord blood. Recipients of non-myeloablative, reduced intensity and myeloablative transplants are eligible.
* Patients who develop acute GVHD after donor lymphocyte infusion (DLI) are eligible.
* There is no specified time window after day 0 of transplant as acute GVHD is only defined by clinical manifestations.
* Patients must have experienced neutrophil engraftment after HSCT as defined by absolute neutrophil counts ≥ 500 / µL × 3 consecutive measurements. Absolute neutrophil count (ANC) should be calculated using the standard formula (Neut + Bands)(WBC × 101).
* The presence of hepatic, upper GI and/or cutaneous acute GVHD is permitted.
* Steroids can be started up to 7 days prior to the administration of natalizumab.
* Age ≥ 18
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study:
* Patients with the entity of Acute/Chronic GVHD overlap syndromes.
* Requiring mechanical ventilation
* Vasopressor requirement
* Concurrent hepatic veno-occlusive disease (VOD) based on clinical examination
* Karnofsky performance status < 30
* Participants may not be receiving any other study agents for at least 7 days prior to enrollment
* Prior use of natalizumab for any reason is not allowed
* Pregnant women are excluded from this study because of the potential teratogenic effects of natalizumab. Because natalizumab enters breast milk, and the effect is unknown in infants, breastfeeding should be discontinued if the mother is treated with natalizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey Cutler, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled subjects with newly diagnosed acute gastrointestinal (GI) graft-versus-host-disease (GVHD) from 2 academic medical centers in the United States. The last patient completed the study in February 2019.
Period: Overall Study
Arm/Group | Natalizumab
Started | 21
Completed | 9
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: Years] | 63 [38 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21
Acute GVHD Staging (Adapted from Glucksberg, H. et al. Transplantation 1974; 18:295) [Count of Participants; unit: Participants] — Skin Stage:
  * 1: Maculopapular rash <25% of body area
  * 2: Maculopapular rash 25-50% of body area
  * 3: Generalized erythroderma
  * 4: Generalized erythroderma with bullous formation and often with desquamation
  Liver Stage:
  * 1: Bilirubin 2.0-3.0 mg/dL
  * 2: Bilirubin 3.1-6.0 mg/dL
  * 3: Bilirubin 6.1-15.0 mg/dL
  * 4: Bilirubin >15.0 mg/dL
  GI Stage:
  * 1: Diarrhea >30 mL/kg or 500 mL/day
  * 2: Diarrhea >60 mL/kg or 1000 mL/day
  * 3: Diarrhea >90 mL/kg or 1500 mL/day
  * 4: Diarrhea >90 mL/kg or 2000 mL/day; or severe abdominal pain with or without ileus
  Participants
    Gastrointestinal Stage 1 | 4
    Gastrointestinal Stage 2 | 5
    Gastrointestinal Stage 3 | 4
    Gastrointestinal Stage 4 | 8
    No liver involvement | 20
    Liver Stage 2 | 1
    No skin involvement | 17
    Skin Stage 2 | 4
Disease Status of Underlying Malignancy at time of Hematopoietic Stem Cell Transplantation (HSCT) [Count of Participants; unit: Participants]
  First Complete Remission | 9
  Second Complete Remission | 5
  Relapsed Disease | 2
  Progressive Disease | 2
  Treatment Failure | 3
Eastern Cooperative Oncology Group (ECOG) Performance Status at HSCT [Count of Participants; unit: Participants]
  00 - Fully Active | 2
  01 - Restricted | 9
  02 - Self Care | 7
  03 - Capable of Limited Self Care | 3
Conditioning Regimen [Count of Participants; unit: Participants]
  Myeloablative | 3
  Non-myeloablative | 18
Donor type [Count of Participants; unit: Participants]
  Matched Unrelated | 15
  Matched Related | 5
  Mismatch Unrelated | 1
Donor source [Count of Participants; unit: Participants]
  Bone marrow and Peripheral Blood Stem Cells | 1
  Peripheral Blood Stem Cells | 20
Acute GVHD Grading (Adapted from Glucksberg, H. et al. Transplantation 1974; 18:295) [Count of Participants; unit: Participants] — * Overall Grade I: Stage 1-2 skin involvement; no liver or GI involvement; ECOG Performance Score 0
  * Overall Grade II: Stage 1-3 skin involvement; Stage 0 liver or GI involvement, ECOG Performance Score 1
  * Overall Grade III: Stage 2-3 skin, liver, or GI involvement; ECOG Performance Score 2
  * Overall Grade IV: Stage 1-4 skin involvement, Stage 2-4 liver or GI involvement, ECOG Performance Score 3
  Participants
    Overall Grade II | 9
    Overall Grade III | 12

OUTCOME MEASURES:

1. Primary Outcome: GVHD-free Survival Rate
Description: Graft-versus-host disease (GVHD) free survival is defined as achieving complete response without death or relapse or requiring secondary immunosuppressive therapy . Proportions are reported descriptively. GVHD-free survival was assessed using the Kaplan-Meier method.
Time Frame: Day 56
Measure: Number; unit: percentage of patients
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
percentage of patients | 33.3

2. Secondary Outcome: Graft-verus-host Disease (GVHD) Response Rate
Description: * Complete Response (CR) is defined as resolution of all signs and symptoms of acute GVHD.
  * Very Good Partial Response (VGPR) is defined by no rash or residual erythematous rash involving less than 25% of the body surface, and total serum bilirubin concentration less than 2 mg/dL or less than 25% of baseline at enrollment and tolerating food or enteral feeding, predominantly formed stools, no overt gastrointestinal bleeding or abdominal cramping, and no more than occasional nausea and vomiting.
  * Partial Response (PR) is defined as an improvement of one stage in one or more organs without progression in any other organ.
  * Non-response (NR) is defined as no reduction in any GVHD organ staging.
  * Progression is defined as either new organ involvement on day +8 or thereafter, or increased organ specific symptoms sufficient to increase the organ stage by one or more or the initiation of an additional GVHD agent.
  * Overall Response Rate (ORR) is the sum of CR, VGPR, and PR.
Time Frame: 28 Days, 56 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
Participants
  Overall Response at Day 28 | 12
  Complete Response at Day 28 | 7
  Very Good Partial Response at Day 28 | 2
  Partial Response at Day 28 | 3
  Non-response/Progression of GVHD at Day 28 | 7
  Overall Response at Day 56 | 11
  Complete Response at Day 56 | 7
  Very Good Partial Response at Day 56 | 2
  Partial Response at Day 56 | 2
  Non-response/Progression of GVHD at Day 56 | 6

3. Secondary Outcome: GI aGVHD Response Rate
Description: Gastrointestinal (GI) acute graft-versus-host disease (GVHD) Response is defined by complete response, very good partial response, or partial response in signs and symptoms of GI aGVHD.
Time Frame: Day 28, Day 56
Measure: Number; unit: percentage of patients
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
percentage of patients
  Overall response rate for GI GVHD at Day 28 | 57
  Overall response rate for GI GVHD at Day 56 | 52

4. Secondary Outcome: Overall Survival (OS) Rate
Description: Overall survival (OS) is defined from the date of natalizumab infusion to death or censored at last clinical evaluation. OS was estimated using the Kaplan-Meier method.
Time Frame: 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
percentage of patients | 43

5. Secondary Outcome: Rate of GVHD Flares
Description: Number of subjects who experienced graft-versus-host disease (GVHD) flares requiring therapy after initial complete response (CR) or partial response (PR) by day 28 after the first dose of Natalizumab.
Time Frame: by Day 28
Measure: Count of Participants; unit: Participants
Groups:
- Natalizumab: Natalizumab-
  * (Day 0 and 28) Fixed dose Intravenous infusion over one hour. 2 hours observation completion of the infusion
  * At 4 weeks, if there has been less than a complete response participants can be treated with a second dose of natalizumab.
  * If participants have no response after one dose, they will be not be given a second dose.
  * Participants who receive a second dose of natalizumab will be evaluated for response at day 56 after first treatment dose administered.
  * Participants will be assessed for response to therapy with natalizumab at day +28, day +56, day +100, day + 180, and day +365.
  * Commercial supplies of Methylprednisolone (or equivalent steroid) will be utilized. The formulation, preparation and route of administration will be as per package insert
  Natalizumab
  Methylprednisolone
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
Participants | 0

6. Secondary Outcome: Percentage Steroid Dose Was Reduced at Day 28, 56, and 100 in Comparison to Steroid Dose at First Administration of Natalizumab.
Description: Median percentage steroid dose was reduced at Day 28, Day 56, and Day 100 in comparison to steroid dose at first administration of Natalizumab.
Time Frame: Day 28, 56, and 100
Measure: Median (Inter-Quartile Range); unit: percentage of steroid dose
Arm/Group | Natalizumab
Number analyzed (Participants) | 21
percentage of steroid dose
  Median reduction in steroid dose at day 28 | 42 [20 to 50]
  Median reduction in steroid dose at day 56 | 71 [60 to 81]
  Median reduction in steroid dose at day 100 | 85 [63 to 93]

ADVERSE EVENTS:
Time Frame: 1 year
Description: All grade 2 related and unexpected and all grade 3 and higher adverse events experienced by participants were collected from the time of the first dose of study treatment, through the study and until the final study visit. Grade 4 skin rash, diarrhea and increased bilirubin were expected adverse events as a result of acute graft-versus-host disease (aGVHD) and did not require reporting. All positive John Cunningham (JC) viral loads required reporting regardless of grade.
Arm/Group | Natalizumab
All-Cause Mortality (participants affected / at risk) | 12/21
Serious Adverse Events (participants affected / at risk) | 8/21
Other Adverse Events (participants affected / at risk) | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natalizumab (N=21)
Hypotension (Cardiac disorders) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1)
Intraparenchymal hemorrhage (Nervous system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Stenotrophomonas bacteremia (Infections and infestations) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
CMV viremia (Infections and infestations) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
C. diff colitis (Infections and infestations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natalizumab (N=21)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Blood and lymphatic system disorders - other (Blood and lymphatic system disorders) | 4 (4)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Cecal infection (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - other (Gastrointestinal disorders) | 4 (4)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Localized edema (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 2 (2)
Hepatobiliary disorders - other (Hepatobiliary disorders) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 3 (3)
Infections and infestations - other (Infections and infestations) | 2 (2)
Small intestine infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Weight loss (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Investigations - other (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (6)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - other (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Nervous system disorders - other (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Renal and urinary disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT02176031/Prot_SAP_000.pdf